CLINICAL TRIAL: NCT00476476
Title: A Phase II Trial of Tarceva (Erlotinib) in Women With Squamous Cell Carcinoma of the Vulvar
Brief Title: Erlotinib in Women With Squamous Cell Carcinoma of the Vulvar
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Neil S. Horowitz, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-174
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-03

CONDITIONS: Squamous Cell Carcinoma
Keywords: Tarceva; erlotinib; squamous cell carcinoma of the vulvar
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib (Experimental): Patients rcvd oral erlotinib 150 mg/day. Cohort 1 pts would have at least 28 days and no more than 42 days of therapy in advance of definitive therapy (surgery or chemoradiation). Cohort 2 pts continued on therapy (28 days per cycle) until disease progression, unacceptable toxicity or withdrawal of consent. Two potential dose reductions were prescribed to 100 and 50 mg/day.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Orally every day for about 4-6 weeks
  Other Names: Tarceva

SUMMARY:
In this research study we are looking to see how vulvar cancer responds to erlotinib therapy. Two distinct patient populations are targeted: women with locally advanced measurable squamous cell carcinoma of the vulva, primary or recurrent, who are candidates for definitive treatment with surgery or chemoradiation (Cohort 1) and women with radiographically measurable distant metastatic cancer either at time of presentation or with recurrence (Cohort 2). Another goal of this study is to learn more about the proteins and genes present in vulvar cancer and how they may affect response to erlotinib. Erlotinib treats cancer by preventing cancer cells from growing and multiplying. It does this by blocking certain proteins that are on the surface of some types of cancer cells. Laboratory tests show that vulvar cancer cells have high levels of these proteins.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

• To determine the clinical efficacy of erlotinib in reducing the size of vulvar squamous cell cancer and /or metastatic lesions.

Secondary

* To determine the safety and tolerability of oral erlotinib.
* To evaluate apoptosis and assess the Ki67, phospho-EGFR, EGFR mutation and EGFR amplification status of the vulvar cancer prior to and after therapy and correlate observed changes with response to therapy.
* To evaluate the impact of medical treatment on the subsequent surgery for vulvar cancer when surgery is chosen as the definitive therapy.

STATISTICAL DESIGN:

This study used a two-stage design to evaluate efficacy of erlotinib based on response determined prior to definitive surgery or chemoradiation (cohort 1) or after every 2 cycles of erlotinib (cohort 2). The null and alternative response rates defined as achieving partial response (PR) or better were 3.5% and 15%. If 1 or more patients enrolled in stage one (n=17 patients) achieved PR or better than accrual would proceed to stage two (n=24 patients). There was 0.55 probability of stopping the trial at stage one if the true OR rate was 3.5%. If 3 or fewer responses were observed by the end of stage two, erlotinib would be deemed ineffective. The significance level of the study design was 0.0495 with a power of 85% to rule out a poor response rate of less than 3.5%.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed measurable squamous cell carcinoma of the vulvar with an assessable lesion on the vulva or measurable metastatic disease. Tumors may be primary or recurrent. Patients must have plans for surgery or definitive treatment with chemotherapy +/-radiation unless they have measurable metastatic disease.
* 18 years of age or older
* No concurrent chemotherapy or radiotherapy
* NO previous chemotherapy or radiotherapy within the preceding 1 month
* ECOG performance status of 0-1

Exclusion Criteria:

* Known hypersensitivity reaction to erlotinib
* Other coexisting malignancies diagnosed within the last 5 years, with the exception of basal cell carcinoma
* Treatment with a non-FDA approved or investigational drug within 30 days
* Persistent toxicities (grade 2 or above) from previous treatment, expect alopecia or lymphedema
* Serum creatinine level greater than CTC grade 2
* Pregnancy or breast feeding
* Severe or uncontrolled systemic disease
* Significant clinical disorder or laboratory finding that makes it potentially unsafe for the subject to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil S. Horowitz, MD, Principal Investigator — Dana-Farber Cancer Institute/Brigham and Women's Hospital
Locations (4):
- United States (4):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island

REFERENCES:
- [Result] Horowitz NS, Olawaiye AB, Borger DR, Growdon WB, Krasner CN, Matulonis UA, Liu JF, Lee J, Brard L, Dizon DS. Phase II trial of erlotinib in women with squamous cell carcinoma of the vulva. Gynecol Oncol. 2012 Oct;127(1):141-6. doi: 10.1016/j.ygyno.2012.06.028. Epub 2012 Jun 26. PMID 22750258

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from February 2007 through July 2011.
Groups:
- Erlotinib-Cohort 1: Patients rcvd oral erlotinib 150 mg/day. Cohort 1 pts would have at least 28 days and no more than 42 days of therapy in advance of definitive therapy (surgery or chemoradiation). Two potential dose reductions were prescribed to 100 and 50 mg/day.
- Erlotinib-Cohort 2: Patients rcvd oral erlotinib 150 mg/day. Cohort 2 pts continued on therapy (28 days per cycle) until disease progression, unacceptable toxicity or withdrawal of consent. Two potential dose reductions were prescribed to 100 and 50 mg/day.
Period: Overall Study
Arm/Group | Erlotinib-Cohort 1 | Erlotinib-Cohort 2
Started | 17 | 24
Response Evaluable | 17 | 23 (One woman was unevaluable due to an allergic reaction that developed after the 2nd dose.)
Completed | 15 | 0 (Treatment was not of fixed duration and thus pts are not considered to have 'Completed' treatment.)
Not Completed | 2 | 24
Not completed — Adverse Event | 2 | 7
Not completed — Progressive Disease | 0 | 17

BASELINE CHARACTERISTICS:
Population: The analysis population is comprised of all enrolled patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib-Cohort 1 | Erlotinib-Cohort 2 | Total
Number analyzed (Participants) | 17 | 24 | 41
Age, Continuous [Mean (Full Range); unit: years] | 75 [58 to 94] | 71.5 [49 to 86] | 73 [49 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 24 | 41
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 24 | 41

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response is defined as achieving complete or partial response.Complete response (CR) for both cohorts was defined as resolution of all identified tumor masses on the vulva or disappearance of all target and non-target lesions with no evidence of new lesions documented by two disease assessments at least 4 weeks apart. For cohort 1 pts, a partial response (PR) was defined as a 30% reduction in the product of all diameters of the vulva tumor/tumors compared to baseline measurements. For cohort 2 pts, PR defined according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) was at least a 30% decrease in the sum of the longest diameter (LD) of all target measurable lesions (baseline sum LD reference).
Time Frame: Assessed prior to definitive surgery or chemoradiation therapy (cohort 1 pts) or after 2 cycles of therapy (cohort 2 pts).
Population: The analysis dataset is comprised of response evaluable patients.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Erlotinib-Cohort 1 | Erlotinib-Cohort 2
Number analyzed (Participants) | 17 | 23
proportion of participants | .35 [.167 to .580] | .22 [.09 to .404]

ADVERSE EVENTS:
Time Frame: Assessed from time of first dose, weekly during treatment and through 30 days post-treatment.
Description: Serious AEs were defined as treatment-related events of grade 3 or higher per CTCAEv3.
  Other AEs were defined as treatment-related events of grades 1 or 2 per CTCAEv3.
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 19/41
Other Adverse Events (participants affected / at risk) | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=41)
Death - disease progression NOS (Investigations) | 2 — Organ System N/A
Hemoglobin (Blood and lymphatic system disorders) | 2
Hearing w/w-o audiogr in monitor prg (Ear and labyrinth disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Infection-other (Infections and infestations) | 1
Bilirubin (Investigations) | 1
Creatinine (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1
Bone, pain (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 1
Perineum, pain (Reproductive system and breast disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=41)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 8
Hematologic-other (Blood and lymphatic system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Endocrine-other (Endocrine disorders) | 1
Dry eye syndrome (Eye disorders) | 1
Eyelid dysfunction (Eye disorders) | 1
Tearing (Eye disorders) | 1
Ocular-other (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 23
Dry mouth (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 7
GI-other (Gastrointestinal disorders) | 3
Abdomen, pain (Gastrointestinal disorders) | 2
Peritoneum, pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 23
Fever w/o neutropenia (General disorders) | 2
Edema limb (General disorders) | 7
Pain-other (General disorders) | 8
Flu-like syndrome (General disorders) | 1
Infection w/ gr3-4 neut, anal/perianal (Infections and infestations) | 1
Infection Gr0-2 neut, lung (Infections and infestations) | 1
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 1
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 3
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 1
Chemoradiation dermatitis (Injury, poisoning and procedural complications) | 1
Leukocytes (Investigations) | 1
Platelets (Investigations) | 1
Weight loss (Investigations) | 3
Alkaline phosphatase (Investigations) | 3
ALT, SGPT (Investigations) | 2
AST, SGOT (Investigations) | 5
Bilirubin (Investigations) | 1
Creatinine (Investigations) | 5
Metabolic/Laboratory-other (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Bicarbonate (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 2
Buttock, pain (Musculoskeletal and connective tissue disorders) | 1
Neck, pain (Musculoskeletal and connective tissue disorders) | 1
Taste disturbance (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 1
Head/headache (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Incontinence urinary (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1
Renal/GU-other (Renal and urinary disorders) | 4
Vagina, hemorrhage (Reproductive system and breast disorders) | 3
Perineum, pain (Reproductive system and breast disorders) | 4
Vagina, pain (Reproductive system and breast disorders) | 3
Vaginal discharge (non-infectious (Reproductive system and breast disorders) | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 12
Alopecia (Skin and subcutaneous tissue disorders) | 6
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 17
Ulceration (Skin and subcutaneous tissue disorders) | 1
Skin-other (Skin and subcutaneous tissue disorders) | 2
Scalp, pain (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Hemorrhage-other (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No